CLINICAL TRIAL: NCT01575457
Title: The Harriet Lane Clinic Healthy Futures Program is to Increase Academic or Workforce Development Success Among Adolescents and Young Adults
Brief Title: Harriet Lane Healthy Futures Program
Acronym: HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Zanvyl and Isabelle Krieger Fund (Other)
Responsible Party: Principal Investigator, Tina L. Cheng, Division Chief, General Pediatrics & Adolescent Medicine, Professor of Pediatrics and Public Health, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 00017226
Record Dates: First submitted 2012-04-08; First posted 2012-04-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Youth Coaching; Future Planning
Keywords: Adolescent Violence Prevention
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The Healthy Futures Program is an interactive, multi-session training program. The intervention participants will participate in College/vocational school, Job, and Career Planning activities with a career coach.
  Interventions: Behavioral: Career Counseling and Motivational Interviewing
- Comparison (Other): The Healthy Futures Program is an interactive, multi-session training program. The comparison group participants will receive newsletters and be invited to participate in college and career planning workshops.
  Interventions: Behavioral: Career Counseling and Motivational Interviewing

INTERVENTIONS:
Behavioral: Career Counseling and Motivational Interviewing — The Healthy Futures Program is an interactive, multi-session training program. There will be participants in 3 different intervention tracks (College/vocational school, Job, and Career Planning). Activities for all three tracks will occur simultaneously. The intervention group will receive the interactive, multi-session training program including newsletters and workshops. Comparison group participants will receive newsletters and be invited to participate in college and career planning workshops.
  Other Names: motivational interviewing; coaching

SUMMARY:
The purpose of the Harriet Lane Clinic Healthy Futures Program is to increase academic or workforce development success among adolescents and young adults. To this end, the Healthy Futures educational intervention includes motivational interviewing and knowledge and skill building activities that will focus on improving educational, vocational, health, and self sufficiency outcomes for youth who attend the Harriet Lane Clinic. Goals of this youth development project include determining what factors are associated with school engagement, parental academic involvement, and future planning.

DETAILED DESCRIPTION:
This is a feasibility study to examine if an intervention in a primary care setting can recruit and retain adolescents and young adults and influence future planning behaviors.

We will address the following research Aims:

1. To assess the feasibility of a career development program provided to low income adolescents and young adults in a pediatric primary care setting.
2. To assess the receptiveness of adolescents and young adults in pediatric primary care setting to future planning interventions.
3. To assess the impact of a career development program in improving educational, workforce, and health attitudes and outcomes for adolescents and young adults.

The Healthy Futures Program is an interactive, multi-session training program. There will be participants in 3 different intervention tracks (College/vocational school, Job, and Career Planning). Tracks are assigned to participants based on interest and age. During the screening process, participants who are 16 years old or older will be asked if they are interested in participating in a program designed to help them apply to college or job training services. Based on their preference, they will be assigned a college or job track. Participants who are 14 and 15 years old will automatically be assigned to the career planning track.

ELIGIBILITY:
Inclusion Criteria:

* The population of interest for this randomized feasibility study are all main-stream (currently or previously enrolled) Baltimore City Public High School 14 to 21 year old attending the Harriet Lane Clinic.

Exclusion Criteria:

* Any student who is currently in a self-contained special education classroom at anytime during the school day will not be invited to participate in the study.
* Students with learning disabilities or physical disabilities that limit their ability to work or read printed materials without assistance will be excluded from the study.
* Lastly, anyone who is not interested in participating in a future planning intervention program will be excluded from the study population.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 202 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Fights in last 30 days | 6 months
  Participants are assessed for fighting behavior 3times (at Baseline, 6months after baseline and 15 months after baseline)

SECONDARY OUTCOMES:
Marijuana use in last 30 days | 6 mo
  Participants are assessed for fighting behavior 3times (at Baseline, 6months after baseline and 15 months after baseline)
Career maturity index | 6 mo
  Participants are assessed for fighting behavior 3times (at Baseline, 6months after baseline and 15 months after baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Harriet Lane Clinic, Baltimore, Maryland, United States